CLINICAL TRIAL: NCT01428557
Title: BREATHE Registry - I Brazilian Registry of Heart Failure
Acronym: BREATHE
Status: Completed | Type: Observational
Sponsor: Hospital do Coracao (Other)
Collaborators: Brazilian Society of Cardiology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 003/2011
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Epidemiology; Evidence-Based Practice
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heart Failure patients (Breathe I): Patients admitted with clinical diagnosis of decompensate heart failure, > 18 years old.
- Heart Failure patients (Breathe Extension): Patients admitted with clinical diagnosis of decompensate heart failure, > 18 years old.

SUMMARY:
The purpose of this study is to evaluate the demographic, clinical, prognostics characteristics of 1,200 patients admitted with clinical diagnosis of decompensate heart failure in a group of 60 hospitals representative in different regions.

DETAILED DESCRIPTION:
Background: Several local registries seek to show an isolated clinical characteristics of patients hospitalized with heart failure (HF) in hospitals and communities in Brazil. Overall, the analysis of these data suggests that there are important differences in etiology, the factors of decompensation, treatment and prognosis of HF patients in different regions.

Objectives: To evaluate the demographic, clinical, prognostics characteristics of 1,200 patients admitted with clinical diagnosis of decompensate heart failure in a group of 60 hospitals representative in different regions. Other specific objectives include describing the in-hospital mortality after admission, to describe the content and the reason for re-admission, to assess adherence to evidence-based guidelines (recommended by guidelines), to measure indicators of quality of care and establish a national registry data to allow for comparison with international records of patients admitted with ADHF.

Methods: Observational cross (record) with longitudinal follow-up where patients admitted to public and private hospitals primarily defined in IC will be studied.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old,
* Boston Criteria > 7,
* patients hospitalized > 24 hours.

Exclusion Criteria:

* myocardial revascularization during last month,
* heart failure due to sepsis,
* acute coronary syndrome with ventricular dysfunction as reason for current hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Public and Private Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 3013 (Actual)
Dates: Start 2011-03; Primary Completion 2019-07 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Total mortality | follow up at 3, 6 and 12 months

SECONDARY OUTCOMES:
Proportion of patients receiving interventions with proven benefit shown by different indicators of quality of care. | follow up at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil